CLINICAL TRIAL: NCT07260214
Title: Effect of Hydrotherapy On Pain, Balance and Quality of Life in Patients With Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Aya Yasser Saber Mahmoud, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPTBSUREC/0305/2325
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrotherapy training (Experimental): This group will consist of seventeen diabetic peripheral neuropathy patients will perform hydrotherapy training for 12 weeks.
  Interventions: Other: Hydrotherapy training
- Land training (Active Comparator): This group will consist of seventeen diabetic peripheral neuropathy patients will do land training for 12 weeks.
  Interventions: Other: Land training

INTERVENTIONS:
Other: Hydrotherapy training — The patients will participate in hydrotherapy sessions three days per week for 12 weeks in a heated swimming pool maintained at 32°C. Each session will include a sequence of activities: relaxation and breath control, balance exercises, gait training, and hydrotherapy cycling.
  Arms: Hydrotherapy training
Other: Land training — The patients do the same exercise of the experimental group on land three days per week for 12 weeks.
  Arms: Land training

SUMMARY:
The current study aims to investigate the effects of hydrotherapy compared to land-based training on patients with diabetic peripheral neuropathy. It will evaluate hydrotherapy's impact on pain relief, sensation improvement, balance, and overall quality of life for these patients.

DETAILED DESCRIPTION:
Hydrotherapy training is a rehabilitative approach proposed for different medical conditions, the hydrotherapy environment facilitates patients with functional limitations, who feel a safer setting and are consequently more motivated to the training. The physical properties of water help to improve patient stability and to allow limbs movements by offloading the body weight and Exerting resistance against the body segments and giving proprioceptive inputs.

Moreover, the warmth of hydrotherapy pool helps muscle relaxation and seems to reduce pain perception, aiming to improve blood circulation so that nutrients can be distributed more smoothly to body tissues, strengthen small muscles, calves, and thighs, as well as address joint mobility limitations often experienced by diabetes mellitus patients.

Several authors evaluated hydrotherapy therapy as possible gait and balance training of neurological patients and demonstrated beneficial effects mostly in Parkinson's disease and stroke. Limited number of studies, even if affected by small sample sizes, made a comparison between hydrotherapy training and on land training. Showing best balance results of the former for the same diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetic peripheral neuropathy due to type 2 diabetes mellitus of both sex Patients must have confirmed diagnosis of diabetic peripheral neuropathy based on clinical symptoms (E.G, numbness, tingling and burning pain) and diagnostic test such as nerve conduction studies
* Chronicity of type 2 diabetes mellitus more than 10 years
* Age range: between 40-65years old
* Stable Blood Glucose Levels HbA1c (≤5.7)
* No active infections or wound

Exclusion Criteria:

* Severe Renal Impairment.
* Uncontrolled cardiovascular diseases
* Pregnancy
* Neurological or musculoskeletal conditions
* Inability to safely enter or exit the pool
* Uncontrolled infections
* Vitamin B12 deficiency.
* Postural hypotension

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Toronto Clinical Neuropathy Score | 12 weeks
  The Toronto Clinical Neuropathy Score (TCNS) is a validated tool for diagnosing and monitoring diabetic sensorimotor peripheral neuropathy (DSPN). It ranges from 0 to 19 points, comprising six points from symptom scores, eight points from lower limb reflexes, and five points from sensory examinations at the toes. The total score categorizes neuropathy severity as follows: 0-5 indicates no neuropathy, 6-8 mild neuropathy, 9-11 moderate neuropathy, and 12 or more indicates severe neuropathy. This scoring system helps clinicians accurately assess neuropathy progression and guide patient management.
McGill pain assessment questionnaire | 12 weeks
  The McGill Pain Questionnaire is a tool used to assess and quantify the severity and characteristics of neuropathic pain, which results from nerve damage or dysfunction. It evaluates pain intensity on a 0-10 scale, where 0 means "no pain" and 10 is the worst possible pain. Patients describe their pain quality using terms like burning, stabbing, electric shock-like, tingling, numbness, and itching. The scoring reflects pain severity, with higher scores indicating more intense pain. This multidimensional tool helps clinicians understand pain characteristics and guide treatment decisions effectively.
Berg balance scale | 12 weeks
  The Berg Balance Scale (BBS) is a widely recognized tool for assessing balance, consisting of 14 items scored on an ordinal scale from 0 to 4, with a total score of 56. Lower scores indicate higher fall risk, where 0 represents the lowest function and 4 the highest. The test typically takes about 20 minutes. Functional levels based on scores include 0-20 indicating ability to walk with a walking aid, 21-40 suggesting walking with assistance, and 41-56 indicating independent walking. The BBS is also used as a fall risk predictor: scores of 41-56 indicate low risk, 21-40 medium risk, and 0-20 high risk.

SECONDARY OUTCOMES:
Diabetes self-Care Activities measurement | 12 weeks
  The Self-Care Activities (SDSCA) scale, developed by Wan Qiaoqin of Peking University, China, will be used to measure the self-care level of patients with diabetic peripheral neuropathy. This scale includes 11 items across six dimensions: general diet, special diet, exercise, blood glucose monitoring, foot care, and medication adherence. Each item will be scored on an eight-point scale from 0 to 7, reflecting the frequency of self-care activities performed by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Ibrahim Abo Elyazed, PhD, Study Chair — Assistant Professor, Beni-Suef University; Reham Ali Mohamed Ali, PhD, Study Director — Lecturer, Beni-Suef University; Ahmed Moheyeldien Hamed, PhD, Study Director — Lecturer, Beni-Suef University
Locations (1):
- Beni-Suef university hospital, Banī Suwayf, Egypt